CLINICAL TRIAL: NCT00903448
Title: Comparison of Prilosec OTC® Versus Prevacid ® for Gastric Acid Suppression
Brief Title: Comparison of Prilosec Over-the-counter (OTC)® Versus Prevacid® for Gastric Acid Suppression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Simon H. Magowan, MD, Procter and Gamble
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2009010
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2010-11-22 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Normal Healthy Subject Population
MeSH Terms: interventions — Omeprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Prilosec OTC
  Interventions: Drug: Prilosec OTC (omeprazole-magnesium)
- B (Active Comparator): Prevacid
  Interventions: Drug: Prevacid

INTERVENTIONS:
Drug: Prilosec OTC (omeprazole-magnesium) — Prilosec OTC (omeprazole-magnesium 20.6 mg) tablet to be taken with a glass of water prior to breakfast
  Arms: A
Drug: Prevacid — Prevacid (15 mg lansoprazole) capsule to be taken with a glass of water prior to breakfast
  Arms: B

SUMMARY:
The objective of this study is to compare Prilosec OTC® to Prevacid® for gastric acid suppression.

ELIGIBILITY:
Inclusion Criteria:

* normal subjects who are age 18-65
* generally healthy
* non-childbearing potential females or those using birth control

Exclusion Criteria:

* history of significant GI disease
* any significant medical illness
* history of hypersensitivity, allergy or intolerance to omeprazole, lansoprazole or other proton pump inhibitors
* currently using GI medications
* GI disorder or surgery leading to impaired drug absorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon H Magowan, MD, Study Director — Procter and Gamble
Locations (1):
- Research Site, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-center, double-blind, randomized, 2-treatment, 3-period cross-over study conducted in forty healthy adult subjects living in the vicinity of the site.
Groups:
- Prilosec OTC Then Prevacid Then Prevacid; Prevacid Then Prilosec OTC Then Prilosec OTC: This study was a 3-period crossover (ABB, BAA). Prilosec OTC (20.6 mg omeprazole magnesium tablet) and Prevacid (15 mg lansoprazole capsule) were administered daily before breakfast.
Period: Period 1: 5 Days Then 10 Day Washout
Arm/Group | Prilosec OTC Then Prevacid Then Prevacid | Prevacid Then Prilosec OTC Then Prilosec OTC
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Period 2: 5 Days Then 10 Day Washout
Arm/Group | Prilosec OTC Then Prevacid Then Prevacid | Prevacid Then Prilosec OTC Then Prilosec OTC
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Period 3: 5 Days
Arm/Group | Prilosec OTC Then Prevacid Then Prevacid | Prevacid Then Prilosec OTC Then Prilosec OTC
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Time That Gastric pH > 4.0 on Day 5
Description: for 24 hours starting Day 5 for each period
Time Frame: 24 hours
Population: This study was a three period, crossover study of 40 subjects entering either treatment sequence ABB or BAA; consequently each subject in the study participated in three periods over which each subject would eventually receive both Prilosec OTC and Prevacid
Measure: Mean (Standard Error); unit: percent time gastric pH exceeds 4.0
Arm/Group | Prilosec OTC Then Prevacid Then Prevacid | Prevacid Then Prilosec OTC Then Prilosec OTC
Number analyzed (Participants) | 40 | 40
percent time gastric pH exceeds 4.0 | 36.8 (3.45) | 45.7 (3.45)
Statistical Analysis 1: Comparison: Prilosec OTC Then Prevacid Then Prevacid vs Prevacid Then Prilosec OTC Then Prilosec OTC; This study enrolled 40 subjects in order to complete a target of at least 30 evaluable subjects. For the purpose of determination of sample size, it was assumed that at least 30 subjects would have complete data for all 3 treatment periods. Assuming the true mean difference in % time that gastric pH > 4.0 between Prilosec OTC and Prevacid was at least 6.5, it was estimated that there would be at least 80% power to detect a treatment difference in 2-sided testing at the 5% significance level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — The least squares treatment means, i.e. adjusted treatment means, and standard errors were computed from the analysis of variance models; Mean Difference (Final Values) = 8.9, Standard Error of Mean 2.1

ADVERSE EVENTS:
Arm/Group | Prilosec OTC Then Prevacid Then Prevacid | Prevacid Then Prilosec OTC Then Prilosec OTC
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 2/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prilosec OTC Then Prevacid Then Prevacid (N=40) | Prevacid Then Prilosec OTC Then Prilosec OTC (N=40)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Skin Disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less